CLINICAL TRIAL: NCT06847854
Title: A Phase I, Multipart, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7497372 Following Intravitreal Administration in Participants With Diabetic Macular Edema (Part 1 Non-Randomized, Open-Label, Multiple Ascending Dose; Part 2 Randomized, Double-Masked)
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of RO7497372 in Participants With Diabetic Macular Edema (DME)
Acronym: Pregonda
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BP44175
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Intervention Model Description: Part 1 is Sequential Assignment. Part 2 is Parallel Assignment.
Who Masked: Participant, Investigator
Masking Description: Part 1: open label; Part 2: double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Multiple Ascending Dose (Experimental): Participants will receive multiple ascending doses of RO7497372, 3 times every 4 weeks (Q4W) as an IVT injection up to Week 8 in the study eye.
  Interventions: Drug: RO7497372
- Part 2: RO7497372 Low Dose (Experimental): Participants will receive 6 doses of RO7497372, low dose, Q4W followed by 3 doses, every eight weeks (Q8W) as an IVT injection up to Week 44 in the study eye.
  Interventions: Drug: RO7497372
- Part 2: RO7497372 High Dose (Experimental): Participants will receive 6 doses of RO7497372, high dose, Q4W followed by 3 doses, Q8W as an IVT injection up to Week 44 in the study eye.
  Interventions: Drug: RO7497372

INTERVENTIONS:
Drug: RO7497372 — RO7497372 will be administered as IVT injection as per the schedule specified in the arms.

SUMMARY:
This study will assess the safety and tolerability of RO7497372 in participants with DME. The study consists of 2 parts. Part 1 will test multiple-ascending doses of RO7497372 after unilateral intravitreal (IVT) administration in participants with DME. The main purpose of Part 1 is to provide data for RO7497372 safety and tolerability, as well as to characterize the ocular and systemic pharmacokinetics (PK), systemic anti-drug antibodies (ADA), and duration of target engagement, i.e., the pharmacodynamics (PD) in aqueous humor (AH) and blood. Part 2 will evaluate the safety, tolerability, PK, and PD of two dose strengths of RO7497372 (low dose and high dose), identified as safe and tolerated in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2), as defined by the world health organization (WHO) and/or American Diabetes Association
* Participant consents to AH collection
* Collection of > 90 microlitres (µL) AH (at each visit required per schedule of activities [SoA]) if deemed feasible and safe by the Investigator.
* Macular thickening secondary to DME involving the center of the fovea with CST >= 325 µm at screening
* Decreased BCVA primarily due to DME with ETDRS score of 78 to 19 letters (both inclusive) at screening
* Adequately clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images
* Diagnosis of non-proliferative DR
* Treatment-naive and Pre-treated participants after washout

Exclusion Criteria:

* Any major illness or major surgical procedure ≤ 4 weeks before Day 1
* Any febrile illness and associated sequelae ≤ 1 week prior to Day 1
* Active cancer ≤ 1 year prior to Day 1
* Cerebral vascular accident (including stroke and transient ischemic attack) or myocardial infarction ≤ 24 weeks prior to Day 1
* HbA1c ≥ 12% at screening
* Any panretinal photocoagulation or macular laser photocoagulation treatment prior to Day 1
* History of vitreoretinal surgery/pars plana vitrectomy
* Any cataract surgery within 12 weeks prior to Day 1 or any planned surgery during the study
* History of any glaucoma surgery including laser glaucoma procedures
* Uncontrolled glaucoma
* Any active intra- or periocular infection on Day 1
* Any active or history of Intraocular inflammation
* Intravitreal treatment with an anti-IL-6 (e.g., vamikibart) or anti-IL-6 receptor treatment at any time
* Any proliferative DR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) | Up to 28 Weeks
Part 2: Number of Participants With Intraocular Inflammation (IOI) AEs as Reported by the Investigator | Baseline to Week 48
Part 2: Number of Participants With Severe or Serious Drug-Related IOI AEs | Baseline to Week 48
  Number of participants with severe or serious drug-related IOI AEs severity will be determined according to the DAIDS toxicity grading scale as reported by the Investigator.
Part 2: Number of Participants With Occlusive Retinal Vasculitis AEs as Reported by the Investigator | Baseline to Week 48

SECONDARY OUTCOMES:
Part 1: Concentration of RO7497372 in Blood | Up to Week 28
Part 1: Concentration of RO7497372 in Aqueous Humor (AH) | Up to Week 28
Part 2: Number of Participants With AEs | Up to 56 weeks
  Number of participants with AEs severity determined according to the DAIDS toxicity grading scale.
Part 2: Number of Participants With Persistent Treatment-induced Anti-drug Antibody (ADAs) | Up to 56 weeks
Part 2: Concentration of RO7497372 in AH | Up to Week 56
Part 2: Concentration of RO7497372 in Plasma | Up to Week 56
Part 2: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score Over Time | From Baseline (Day 1) up to Week 56
  BCVA will be measured via Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters using a set of three Precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity (VA) examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicates improvement in VA.
Part 2: Absolute Value of BCVA Score Over Time | Up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicates improvement in VA.
Part 2: Percentage of Participants Gaining ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | Up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicates improvement in VA.
Part 2: Percentage of Participants Avoiding a Loss of ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | Up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three Precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicates improvement in VA.
Part 2: Change From Baseline in Central Subfield Thickness (CST) Over Time | From Baseline (Day 1) up to Week 56
  CST is defined as the average thickness of the central 1-mm circle of the ETDRS grid centered to the fovea measured between the internal limiting membrane and the Bruch's membrane. CST will be determined by CRC evaluation of SD-OCT images.
Part 2: Absolute Value of CST Over Time | Up to Week 56
  CST is defined as the average thickness of the central 1-mm circle of the ETDRS grid centered to the fovea measured between the internal limiting membrane and the Bruch's membrane. CST will be determined by CRC evaluation of SD-OCT images.
Part 2: Percentage of Participants With Absence of DME Over Time | Up to Week 56
  Absence of DME is defined as CST < 325 micrometre (μm) by spectral domain optical coherence tomography (SD-OCT).
Part 2: Percentage of Participants With Absence of Intraretinal Fluid and/or Subretinal Fluid Over Time | Up to Week 56
  Presence of intraretinal and subretinal fluid will be determined by CRC evaluation of SD -OCT images.
Part 2: Percentage of Participants With ≥ 2-step Diabetic Retinopathy Severity Scale (DRSS) Improvement From Baseline on the ETDRS DRSS Over Time | Up to Week 56
  The DRSS will be graded according to ETDRS grading schedules from report 18 JOVS, February 1998, Vol. 39, No. 2. ETDRS DRSS is 13 step scale which measures severity of diabetic retinopathy (DR). The DRSS scores vary from 10 (DR absent) to 90 (ungradable proliferative diabetic retinopathy(PDR)). Higher levels indicate higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (37):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Consultants of AZ, Ltd, Peoria, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Arkansas Retina Research, Little Rock, Arkansas
  - Global Research Management, Glendale, California
  - Retinal Consultants Medical Group, Modesto, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Florida Eye Associates, Melbourne, Florida
  - Medeye Associates, Miami, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Center for Retina and Macula Disease, Winter Haven, Florida
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Retina Consultants Minnesota, Saint Louis Park, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Ross Eye Institute, Buffalo, New York
  - Retina Associates of NY, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Verum Research LLC, Eugene, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Austin Clinical Research LLC, Austin, Texas
  - Brown Retina Institute, Schertz, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Salt Lake Retina, West Jordan, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- Emanuelli Research and Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No